CLINICAL TRIAL: NCT06114264
Title: Multimodal Intervention to Improve Pain and Health in Patients With Non-specific Chronic Low Back Pain: the HEALTHY BACK Project
Brief Title: Multimodal Intervention in Patients With Non-specific Chronic Low Back Pain: the HEALTHY BACK Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBS Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Víctor Segura Jiménez, Principal Investigator, IBS Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iBSGranada
Record Dates: First submitted 2023-10-10; First posted 2023-11-02 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pain, Chronic; Neurologic Manifestations; Back Pain; Low Back Pain; Behavior, Health
Keywords: exercise; behaviour change; education; mindfulness; pain; strength
MeSH Terms: conditions — Chronic Pain; Neurologic Manifestations; Back Pain; Low Back Pain; Health Behavior; Motor Activity; Pain | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): This group will not receive any treatment during the intervention period.
  Interventions: Other: Control group
- Multimodal + Resistance Program (Experimental): Multimodal program including exercise program 2 days / week (45 minutes per session) during a period of 8 weeks + Behaviour change program daily /24 hours via a wrist-worn activity prompting device during a period of 8 weeks + Education program 2 days / week (1.5 hour per session, except the final session lasting 2 hours) during a period of 3 weeks + Mindfulness intervention 1 day / week (2.5 hour per session) during a period of 8 weeks, and will continue with an extended exercise program (functional resistance training) additionally 3 days / week (50 minutes per session) during 8 weeks.
  Interventions: Behavioral: Multimodal + Resistance Programs

INTERVENTIONS:
Behavioral: Multimodal + Resistance Programs — Exercise: will focus on working the all body by performing functional tasks. Behaviour change: An 'idle alert' of the wrist-worn activity prompter will be set to vibrate after 45 min without movement. Participants will be encouraged to take a 1-2 min activity break.
  Education: The basic contents will explain to the patient the main mechanism of chronic pain (pain as a protective system, consequences, etc).
  The Mindfulness Based Stress Reduction (MBSR) program will strictly follow the protocol developed by Jon Kabat Zinn. Each session will include three activities: the presentation of a topic, moments of dialogue and exploration in group and a Mindfulness practice.
  Resistance functional exercises will replicate functional movements, such as standing from a bed, carrying bags, picking up groceries from the ground, etc.
  Arms: Multimodal + Resistance Program
Other: Control group — No experimental intervention. The group will receive the same multimodal intervention as the experimental group when the experimental period is over.
  Arms: Control Group

SUMMARY:
Low back pain is one of the most common health problems seen in the primary care. Chronic low back pain is localized between the inferior limit of the ribs and the sacral region, and persist more than 12 weeks. In most cases, it is attributed to a non-specific cause and classified as non-specific chronic low back pain (NSCLBP). No previous study has included a multimodal supervised program in patients with NSCLBP. The primary aim of this study is to determine the effectiveness of exercise + behaviour change + education + mindfulness programs (intervention 1) and an intervention including intervention 1 following functional resistance training (Intervention 2) on endogenous pain modulation, disability, muscle strength/endurance, quality of life, gait parameters, levels of physical activity, sedentary behaviour and psychological health in patients with NSCLBP.

ELIGIBILITY:
Inclusion Criteria:

* Be previously diagnosed with NSCLBP pain by a healthcare professional according to the criteria established by O'Sullivan et al1.
* Intend to participate in the intervention and perform all the tests included in the study.
* Able to read and understand informed consent, as well as the objective of the study.
* Able to walk and move without outside help.
* Able to communicate without problems.

Exclusion Criteria:

* Be under 20 years or over 65 years old.
* Having acute or terminal illness.
* Having medical prescription that prevents the performance of the tests.
* Having injury or circumstance that makes it impossible to perform the tests correctly.
* Having other physical or mental illness that prevents participating in the intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Conditioned Pain Modulation (CPM) in the lower back at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured using the sphygmomanometer on the upper arm contralateral to the most painful lumbar side.
Change from baseline Conditioned Pain Modulation (CPM) in the lower back at 3.5 months | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be measured using the sphygmomanometer on the upper arm contralateral to the most painful lumbar side.
Change from baseline Conditioned Pain Modulation (CPM) in the lower back at 5 months | Change from baseline at 5 months (Retest minus Pretest)
  It will be measured using the sphygmomanometer on the upper arm contralateral to the most painful lumbar side.
Change from baseline Temporal Sumation of Pain (TSP) in the lower back at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Temporal Sumation of Pain (TSP) in the lower back at 3.5 months | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Temporal Sumation of Pain (TSP) in the lower back at 5 months | Change from baseline at 5 months (Posttest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Pressure pain threshold (PPT) in the lower back at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Pressure pain threshold (PPT) in the lower back at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).
Change from baseline Pressure pain threshold (PPT) in the lower back at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be measured using a hand-held standard pressure algometer (FPK 20, Wagner Instruments, Greenwich, CT, USA).

SECONDARY OUTCOMES:
Change from baseline Disability due to pain at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be assessed with the Oswestry low back pain scale. The total score will be calculated summing the value of the 10 items and represented as percentage (%), where 0-20% means minimum functional limitation; 20%-40% moderate functional limitation; 40%-60% intense functional limitation; 60%-80% disability and more than 80% maximum functional limitation.
Change from baseline Disability due to pain at 3.5 months | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be assessed with the Oswestry low back pain scale. The total score will be calculated summing the value of the 10 items and represented as percentage (%), where 0-20% means minimum functional limitation; 20%-40% moderate functional limitation; 40%-60% intense functional limitation; 60%-80% disability and more than 80% maximum functional limitation.
Change from baseline Disability due to pain at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be assessed with the Oswestry low back pain scale. The total score will be calculated summing the value of the 10 items and represented as percentage (%), where 0-20% means minimum functional limitation; 20%-40% moderate functional limitation; 40%-60% intense functional limitation; 60%-80% disability and more than 80% maximum functional limitation.
Change from baseline Pain intensity at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  Patients will be instructed to indicate the intensity of pain they felt on a valid and reliable 10 cm long straight line marked with a score from 0 to 10.
Change from baseline Pain intensity at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Patients will be instructed to indicate the intensity of pain they felt on a valid and reliable 10 cm long straight line marked with a score from 0 to 10.
Change from baseline Pain intensity at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Patients will be instructed to indicate the intensity of pain they felt on a valid and reliable 10 cm long straight line marked with a score from 0 to 10.
Change from baseline physical activity and sedentary time at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  They will be recorded through GT3X+ Accelerometer (Actigraph, Inc., Fort Walton Beach, FL, USA).
Change from baseline physical activity and sedentary time at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  They will be recorded through GT3X+ Accelerometer (Actigraph, Inc., Fort Walton Beach, FL, USA).
Change from baseline physical activity and sedentary time at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  They will be recorded through GT3X+ Accelerometer (Actigraph, Inc., Fort Walton Beach, FL, USA).
Change from baseline Gait parameters at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, gait speed (m/s) will be calculated using Optogait platform.
Change from baseline Gait parameters at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, gait speed (m/s) will be calculated using Optogait platform.
Change from baseline Gait parameters at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Spatiotemporal gait parameters such as, gait speed (m/s) will be calculated using Optogait platform.
Change from baseline Gait parameters at 2 months control and intervention group 1 | Change from baseline at 2 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, stride length (cm) will be calculated using Optogait platform.
Change from baseline Gait parameters at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, stride length (cm) will be calculated using Optogait platform.
Change from baseline Gait parameters at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Spatiotemporal gait parameters such as, stride length (cm) will be calculated using Optogait platform.
Change from baseline Gait parameters at 2 months control and intervention group 1 | Change from baseline at 2 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, load response (gr/cm^2) will be calculated using Optogait platform.
Change from baseline Gait parameters at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, load response (gr/cm^2) will be calculated using Optogait platform.
Change from baseline Gait parameters at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Spatiotemporal gait parameters such as, load response (gr/cm^2) will be calculated using Optogait platform.
Change from baseline Gait parameters at 2 months control and intervention group 1 | Change from baseline at 2 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, double support (s) will be calculated using Optogait platform.
Change from baseline Gait parameters at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Spatiotemporal gait parameters such as, double support (s) will be calculated using Optogait platform.
Change from baseline Gait parameters at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Spatiotemporal gait parameters such as, double support (s) will be calculated using Optogait platform.
Change from baseline Fat percentage at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  Will be measured by bioelectrical impedance analysis (InBody R20, Biospace)
Change from baseline Fat percentage at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Will be measured by bioelectrical impedance analysis (InBody R20, Biospace)
Change from baseline Fat percentage at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Will be measured by bioelectrical impedance analysis (InBody R20, Biospace)
Change from baseline weight (kg) and height (cm) to report BMI in kg/m^2 at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  They will be measured by bioelectrical impedance analysis (InBody R20, Biospace) and height rod (Seca 22).
Change from baseline weight (kg) and height (cm) to report BMI in kg/m^2 at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  They will be measured by bioelectrical impedance analysis (InBody R20, Biospace) and height rod (Seca 22).
Change from baseline weight (kg) and height (cm) to report BMI in kg/m^2 at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  They will be measured by bioelectrical impedance analysis (InBody R20, Biospace) and height rod (Seca 22).
Change from baseline Health-related quality of life at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  Will be assessed with the Short-Form Health Survey (SF-36). It contains 36 items grouped into 8 dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health. The scores range from 0 to 100 in every dimension, where higher scores indicate better health.
Change from baseline Health-related quality of life at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Will be assessed with the Short-Form Health Survey (SF-36). It contains 36 items grouped into 8 dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health. The scores range from 0 to 100 in every dimension, where higher scores indicate better health.
Change from baseline Health-related quality of life at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Will be assessed with the Short-Form Health Survey (SF-36). It contains 36 items grouped into 8 dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health. The scores range from 0 to 100 in every dimension, where higher scores indicate better health.
Change from baseline Central sensitization at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  The Central Sensitisation Inventory will be used. It is a self-report questionnaire designed to identify patients who have symptoms that may be related to central sensitisation. It presents 25 questions and the patient scores each answer on a scale of 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation.
Change from baseline Central sensitization at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  The Central Sensitisation Inventory will be used. It is a self-report questionnaire designed to identify patients who have symptoms that may be related to central sensitisation. It presents 25 questions and the patient scores each answer on a scale of 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation.
Change from baseline Central sensitization at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  The Central Sensitisation Inventory will be used. It is a self-report questionnaire designed to identify patients who have symptoms that may be related to central sensitisation. It presents 25 questions and the patient scores each answer on a scale of 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation.
Change from baseline Pain Catastrophyzing at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  The Pain Catastrophizing Scale will be used to assess painful experiences and thoughts or feelings about pain. It contains 13 items on a 5-point scale. Higher score represents a more negative appraisal of pain.
Change from baseline Pain Catastrophyzing at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  The Pain Catastrophizing Scale will be used to assess painful experiences and thoughts or feelings about pain. It contains 13 items on a 5-point scale. Higher score represents a more negative appraisal of pain.
Change from baseline Pain Catastrophyzing at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  The Pain Catastrophizing Scale will be used to assess painful experiences and thoughts or feelings about pain. It contains 13 items on a 5-point scale. Higher score represents a more negative appraisal of pain.
Change from baseline Depression severity at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  The Beck Depression Inventory-II will be used. It contains 21 items and the range of score is 0-63 with higher values indicating greater depression.
Change from baseline Depression severity at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  The Beck Depression Inventory-II will be used. It contains 21 items and the range of score is 0-63 with higher values indicating greater depression.
Change from baseline Depression severity at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  The Beck Depression Inventory-II will be used. It contains 21 items and the range of score is 0-63 with higher values indicating greater depression.
Change from baseline Anxiety state at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  The State Trait Anxiety Inventory-I will be used to assess anxiety state (i.e., the level of current anxiety). It is a 20-item self-administered questionnaire and the range of score is 20-80, with higher score indicating a greater anxiety state.
Change from baseline Anxiety state at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  The State Trait Anxiety Inventory-I will be used to assess anxiety state (i.e., the level of current anxiety). It is a 20-item self-administered questionnaire and the range of score is 20-80, with higher score indicating a greater anxiety state.
Change from baseline Anxiety state at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  The State Trait Anxiety Inventory-I will be used to assess anxiety state (i.e., the level of current anxiety). It is a 20-item self-administered questionnaire and the range of score is 20-80, with higher score indicating a greater anxiety state.
Change from baseline Sleep duration and quality at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be assessed with the Pittsburgh Sleep Quality Index. It is composed of 19 questions, with four-point Likert scales (0-3), addressing seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The sleep quality global score is the sum of all components. Higher scores indicate worse sleep quality.
Change from baseline Sleep duration and quality at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be assessed with the Pittsburgh Sleep Quality Index. It is composed of 19 questions, with four-point Likert scales (0-3), addressing seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The sleep quality global score is the sum of all components. Higher scores indicate worse sleep quality.
Change from baseline Sleep duration and quality at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be assessed with the Pittsburgh Sleep Quality Index. It is composed of 19 questions, with four-point Likert scales (0-3), addressing seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The sleep quality global score is the sum of all components. Higher scores indicate worse sleep quality.
Change from baseline Haemostasis at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be carried out with a blood draw. The Haemostasis will include prothrombin time (seconds)
Change from baseline Haemostasis at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be carried out with a blood draw. The Haemostasis will include prothrombin time (seconds)
Change from baseline Haemostasis at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be carried out with a blood draw. The Haemostasis will include prothrombin time (seconds)
Change from baseline Specific Proteins at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be carried out with a blood draw. The specific proteins will be reactive protein C (mg/L)
Change from baseline Specific Proteins at 3.5 months | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be carried out with a blood draw. The specific proteins will be reactive protein C (mg/L)
Change from baseline Specific Proteins at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be carried out with a blood draw. The specific proteins will be reactive protein C (mg/L)
Change from baseline Specific Proteins at 2 months control and intervention group 1 | Change from baseline at 2 months control and intervention group 1 (Posttest minus Pretest)
  It will be carried out with a blood draw. The specific proteins will be interleukin 6 (pg/mL)
Change from baseline Specific Proteins at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be carried out with a blood draw. The specific proteins will be interleukin 6 (pg/mL)
Change from baseline Specific Proteins at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be carried out with a blood draw. The specific proteins will be interleukin 6 (pg/mL)
Change from baseline Hormones at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be carried out with a blood draw. The Hormones will be cortisol (μg/dL).
Change from baseline Hormones at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be carried out with a blood draw. The Hormones will be cortisol (μg/dL).
Change from baseline Hormones at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be carried out with a blood draw. The Hormones will be cortisol (μg/dL).
Change from baseline Vitamin D-25OH at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  Vitamin D-25OH (ng/mL) will be carried out with a blood draw.
Change from baseline Vitamin D-25OH at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  Vitamin D-25OH (ng/mL) will be carried out with a blood draw.
Change from baseline Vitamin D-25OH at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  Vitamin D-25OH (ng/mL) will be carried out with a blood draw.
Change from baseline Immunology at 2 months | Change from baseline at 2 months (Posttest minus Pretest)
  It will be carried out with a blood draw. The General Immunology will include C3 and C4 complement (mg/dL)
Change from baseline Immunology at 3.5 months control and intervention group 1 | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be carried out with a blood draw. The General Immunology will include C3 and C4 complement (mg/dL)
Change from baseline Immunology at 5 months control and intervention group 1 | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be carried out with a blood draw. The General Immunology will include C3 and C4 complement (mg/dL)
Change from baseline Muscular fitness at 5 months control and intervention group 1: isometric and isokinetic trunk flexor and extensor strength | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will me measured with the electromechanic functional dynamometer (DYNASYSTEM, Granada, Spain)
Change from baseline Muscular fitness at 3.5 months control and intervention group 1: isometric and isokinetic trunk flexor and extensor strength | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will me measured with the electromechanic functional dynamometer (DYNASYSTEM, Granada, Spain)
Change from baseline Muscular fitness at 2 months: isometric and isokinetic trunk flexor and extensor endurance/strength | Change from baseline at 2 months (Posttest minus Pretest)
  It will me measured with the electromechanic functional dynamometer (DYNASYSTEM, Granada, Spain)
Change from baseline Muscular fitness at 5 months control and intervention group 1: cardio-respiratory fitness | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be measured with the YMCA 3 minutes step test
Change from baseline Muscular fitness at 3.5 months control and intervention group 1: cardio-respiratory fitness | Change from baseline at 3.5 months control and intervention group 1 (Posttest minus Pretest)
  It will be measured with the YMCA 3 minutes step test
Change from baseline Muscular fitness at 2 months: cardio-respiratory fitness | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured with the YMCA 3 minutes step test
Change from baseline Muscular fitness at 5 months control and intervention group 1: upper body strength | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be measured with the handgrip strength test (TKK 5101 Grip-D dynamometer; Takei Scientific Instruments Co., Ltd., Tokyo, Japan).
Change from baseline Muscular fitness at 3.5 months: upper body strength | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be measured with the handgrip strength test (TKK 5101 Grip-D dynamometer; Takei Scientific Instruments Co., Ltd., Tokyo, Japan).
Change from baseline Muscular fitness at 2 months: upper body strength | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured with the handgrip strength test (TKK 5101 Grip-D dynamometer; Takei Scientific Instruments Co., Ltd., Tokyo, Japan).
Change from baseline Muscular fitness at 5 months control and intervention group 1: lower body endurance | Change from baseline at 5 months control and intervention group 1 (Retest minus Pretest)
  It will be measured by the 30s chair stand test.
Change from baseline Muscular fitness at 3.5 months: lower body endurance | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be measured by the 30s chair stand test.
Change from baseline Muscular fitness at 2 months: lower body endurance | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured by the 30s chair stand test.
Change from baseline Muscular fitness at 2 months: The trunk muscle endurance | Change from baseline at 2 months (Posttest minus Pretest)
  It will be measured with the Biering-Sørensen test (seconds per minute) and the prone bridging test (seconds per minute).
Change from baseline Muscular fitness at 3.5 months: The trunk muscle endurance | Change from baseline at 3.5 months (Posttest minus Pretest)
  It will be measured with the Biering-Sørensen test (seconds per minute) and the prone bridging test (seconds per minute).
Change from baseline Muscular fitness at 5 months: The trunk muscle endurance | Change from baseline at 5 months (Retest minus Pretest)
  It will be measured with the Biering-Sørensen test (seconds per minute) and the prone bridging test (seconds per minute).

CONTACTS AND LOCATIONS:
Locations (1):
- iBS.Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsiarleston G, Lopez-Fernandez MD, Pavon-Munoz R, Aguilera-Garcia I, Lopez-Corchon M, Delgado-Fernandez M, Castellote-Caballero MY, Donoso B, Mesa-Ruiz AM, Pozuelo-Calvo R, Rios-Ortiz AM, Alvarez-Corral G, Marin-Jimenez N, Martinez-Garcia D, Chirosa Rios IJ, Segura-Jimenez V. Multimodal intervention based on physical exercise, mindfulness, behaviour change and education to improve pain and health in patients with chronic primary low back pain: a study protocol of the HEALTHYBACK randomised controlled trial. BMJ Open Sport Exerc Med. 2024 Nov 21;10(4):e002188. doi: 10.1136/bmjsem-2024-002188. eCollection 2024. PMID 39610994